CLINICAL TRIAL: NCT00110136
Title: A Phase II Study of St. John's Wort for the Treatment of Hot Flashes in Women With a History of Breast Cancer
Brief Title: St. John's Wort in Relieving Hot Flashes in Postmenopausal Women With Non-Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped due to concerns about interaction between St. John's wort and Tamoxifen.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REBACCCWFU 98301; U10CA081851 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; breast cancer in situ; ductal breast carcinoma in situ; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Hypericum extract LI 160

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- St. John's Wort (Experimental): Patient given one 300mg St. John's Wort tablet three times per day
  Interventions: Drug: St. John's Wort

INTERVENTIONS:
Drug: St. John's Wort — St. John's Wort 300mg tablet three times per day

SUMMARY:
RATIONALE: St. John's wort may help relieve hot flashes in women with breast cancer.

PURPOSE: This phase II trial is studying how well St. John's wort works in relieving hot flashes in women with non-metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of Hypericum perforatum (St. John's wort) in alleviating hot flashes, in terms of hot flash frequency, score, and duration and disruption of daily activities caused by hot flashes, in postmenopausal women with non-metastatic breast cancer.
* Determine hot flash changes over 4 weeks in patients treated with this drug.

Secondary

* Determine the toxicity of this drug in these patients.
* Determine the effect of Hypericum perforatum (St. John's wort) on serum tamoxifen levels in women receiving tamoxifen therapy.
* Determine the effect of Hypericum perforatum (St. John's wort) on general health-related quality of life and mood at 2 and 4 weeks relative to baseline, and during the 2 week post-treatment phase in these patients.
* To evaluate changes in average weekly hot flush scores and duration over course of study.

OUTLINE: This is a multicenter study.

Patients receive oral Hypericum perforatum (St. John's wort) three times daily for 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete a daily diary of the frequency, severity, and duration of their hot flashes, and complete quality of life and mood assessments every 2 weeks during study treatment and continuing weekly for 2 weeks after completion of study treatment.

Patients receiving tamoxifen will have blood tests to measure serum tamoxifen levels at baseline, 2, 4, and 6 weeks.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Noninvasive ductal carcinoma in situ
  * Localized breast cancer

    * Stage 0-IIIB disease
  * Locally recurrent breast cancer that is post-treatment AND disease-free for ≥ 2 years
* Experiencing ≥ 3 hot flashes per day (≥ 21 per week), defined by sweating, flushing, sensation of warmth, night sweats, and/or rapid heart beat of sufficient severity that the patient desires therapeutic intervention
* Normal mammogram within the past 10 months
* Hormone receptor status:

  * Not specified

INCLUSION CRITERIA:

Age

* 18 and over

Sex

* Female

Menopausal status

* Post-menopausal (i.e., no menstrual periods ≥ 12 months or surgical menopause)

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2 mg/dL
* SGOT ≤ 2 times normal

Renal

* Not specified

EXCLUSION CRITERIA:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of intolerance to St. John's wort

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent cytotoxic chemotherapy

Endocrine therapy

* No concurrent selective estrogen-receptor modulators or aromatase inhibitors (e.g., anastrozole, letrozole, or exemestane) allowed

  * Concurrent tamoxifen allowed
* No concurrent estrogen, progestational agents, or androgens for the alleviation of hot flashes
* No concurrent corticosteroids

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 14 days since prior Hypericum perforatum (St. John's wort), monoamine oxidase inhibitors, selective serotonin reuptake inhibitors (e.g., sertraline, paroxetine, or fluoxetine) or selective norepinephrine reuptake inhibitors (e.g., venlafaxine)
* No concurrent use of any of the following:

  * Antidepressants
  * Theophylline
  * Warfarin, unless for central line prophylaxis
  * Protease inhibitors for AIDS
  * Digoxin
  * Cyclosporine
  * Benzodiazepines (e.g., diazepam or alprazolam)
  * Calcium-channel blockers (e.g., diltiazem or nifedipine)
  * Coenzyme A reductase inhibitors for serum cholesterol reduction
  * Macrolide antibiotics (e.g., azithromycin, erythromycin, or clarithromycin)
  * Griseofulvin
  * Phenobarbital
  * Phenytoin
  * Rifampin
  * Rifabutin
  * Grapefruit juice
  * Other naturopathic or herbal products
  * Ketoconazole
  * Fluconazole
  * Itraconazole
  * Rifabutin
* No other concurrent medications for the alleviation of hot flashes (e.g., clonidine or bellamine)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-03-16 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2008-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Naughton, PhD, Study Chair — Wake Forest University Health Sciences
Locations (19):
- United States (19):
  - Helen F. Graham Cancer Center at Christiana Hospital, Newark, Delaware
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Hugh Chatham Memorial Hospital, Elkin, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | St. John's Wort
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All registered participants are used in the analysis.
Arm/Group | St. John's Wort
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (7.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 9
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Effect of St. John's Wort on Hot Flash Frequency as Recorded in a Daily Hot Flash Diary From Baseline to 4 Weeks
Description: Primary objective was to assess the change in hot flashes over a four week period in patients given St. John's Wort
Time Frame: Baseline and four weeks
Population: All registered participants
Measure: Mean (Standard Deviation); unit: number of occurrences
Arm/Group | St. John's Wort
Number analyzed (Participants) | 9
number of occurrences
  Baseline | 7.8 (5.3)
  Four Weeks | 7.0 (5.3)
Statistical Analysis 1: Comparison: St. John's Wort; Analysis of the change in hot flash frequency from baseline to four weeks; null hypothesis is no change; Test type: Superiority or Other; p = 0.2629, paired t-test — Paired t-test; no adjustments for multiple comparisons; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-2.36 to 0.74], Standard Deviation 2.02 — The difference is post minus pre so negative values represents fewer hot flashes after treatment

2. Secondary Outcome: Effect of St. John's Wort on Hot Flash Score as Recorded in a Daily Hot Flash Diary From Baseline to 4 Weeks
Description: The hot flash score is calculated as the frequency of hot flashes times the severity of the hot flashes averaged over a week.
  Frequency is the number of hot flashes in a day. Severity is coded 0=None, 1=Mild, 2=Moderate, and 3=Severe. Score for each day is frequency times severity. Weekly score is averaged over seven days.
  Score ranges from 0 to infinity
  Lower scores are better.
Time Frame: Baseline and four weeks
Population: All registered participants
Measure: Mean (Standard Deviation); unit: frequency times severity
Arm/Group | St. John's Wort
Number analyzed (Participants) | 9
frequency times severity
  Baseline | 19.4 (17.5)
  Four Weeks | 15.0 (17.3)
Statistical Analysis 1: Comparison: St. John's Wort; Assessment of the change in the hot flash score over time; Test type: Superiority or Other; p = 0.1365, paired t-test — Paired t-test; unadjusted for multiple comparisons; Mean Difference (Final Values) = -4.37, 95% CI 2-sided [-10.45 to 1.72], Standard Deviation 7.91 — Difference in hot flash score is post minus pre so a negative value represents a decrease in the frequency and/or severity of the hot flashes

3. Secondary Outcome: Estimation of Toxicities While on St. John's Wort
Description: Toxicities are quantified using the standard NCI toxicity criteria. The outcome is the percentage of participants who experience one or more toxicities. More detailed information on toxicities is found in the adverse events section.
Time Frame: Six weeks following baseline (four weeks of active treatment and two weeks of follow-up)
Population: All registered participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | St. John's Wort
Number analyzed (Participants) | 9
percentage of participants | 66.67 [29.93 to 92.51]

4. Secondary Outcome: Effect of St. John's Wort on Quality of Life (MCS)
Description: Quality of life was measured by the SF12 (MCS and PCS subscales). First we'll summarize the MCS.
  SF-12 is the short form Health Survey (a short version of the SF-36) developed for the Medical Outcomes Study. It is managed by QualityMetric.
  MCS is the mental health component of the SF-12. A normal population has a mean of 50 and a SD of 10. Higher numbers represent better mental health.
  The range is 0 to 100.
  Higher scores represent better mental health.
Time Frame: Baseline and four weeks
Population: All registered participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | St. John's Wort
Number analyzed (Participants) | 9
units on a scale
  Baseline | 53.3 (7.5)
  Four Weeks | 53.8 (4.0)
Statistical Analysis 1: Comparison: St. John's Wort; Assess the change in MCS from baseline to four weeks in patients receiving St. John's wort; Test type: Superiority or Other; p = 0.8320, paired t-test — Paired t-test; unadjusted for multiple comparisons; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [-4.84 to 5.92], Standard Deviation 7.00 — This is the change in MCS from baseline to four weeks (post minus pre) so values greater than zero reflect improvement in QOL

5. Secondary Outcome: Effect of St. John's Wort on Quality of Life (PCS)
Description: Quality of life was measured by the SF12 (MCS and PCS subscales). Now we'll summarize the PCS.
  SF-12 is the short form Health Survey (a short version of the SF-36) developed for the Medical Outcomes Study. It is managed by QualityMetric.
  PCS is the physical health component of the SF-12. Normal population has a mean of 50 and a SD of 10. Higher scores reflect better physical health.
  The range is 0 to 100.
  Higher scores represent better mental health.
Time Frame: Baseline and four weeks
Population: All registered participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | St. John's Wort
Number analyzed (Participants) | 9
units on a scale
  Baseline | 47.4 (12.6)
  Four Weeks | 47.4 (9.6)
Statistical Analysis 1: Comparison: St. John's Wort; Assess the change in PCS from baseline to four weeks; null hypothesis is no change; Test type: Superiority or Other; p = 0.9995, paired t-test — Paired t-test on the change in PCS from baseline to four weeks; unadjusted for multiple comparisons; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-5.71 to 5.71], Standard Deviation 7.43 — This is the change in PCS from baseline to four weeks (post minus pre), so positive numbers represent improvement in QOL

6. Secondary Outcome: Mood is Measured by the POMS Short Form.
Description: POMS stands for the Profile of Mood States This is a short version of the POMS (17 questions).
  Each question is scored on a 0 to 4 scale. The POMS score is the sum of the responses to the 17 questions. Responses to some questions have been reversed to make higher responses better.
  The range is 0 to 68.
  Higher scores represent better overall mood.
Time Frame: Baseline and four weeks
Population: All registered participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- St. John's Wort: Patients given one 300mg St. John's Wort tablet three times per day
  St. John's Wort: St. John's Wort 300mg tablet three times per day
Arm/Group | St. John's Wort
Number analyzed (Participants) | 9
units on a scale
  Baseline | 51.7 (8.4)
  Four Weeks | 56.1 (3.4)
Statistical Analysis 1: Comparison: St. John's Wort; Assess the change in mood from baseline to four weeks. Null hypothesis is no change; Test type: Superiority or Other; p = 0.1042, paired t-test — Paired t-test; unadjusted for multiple comparisons; Mean Difference (Final Values) = 4.35, 95% CI 2-sided [-1.12 to 9.822], Standard Deviation 7.12 — This is the change in mood from baseline to four weeks (post minus pre). Mood is scored so that higher numbers represent better mood so positive changes represent an improvement in mood

ADVERSE EVENTS:
Time Frame: Ten weeks
Arm/Group | St. John's Wort
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | St. John's Wort (N=9)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dizziness (Nervous system disorders) | 3 (4)
Dry Mouth (Gastrointestinal disorders) | 4 (9)
Fatigue (General disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (3)
Hot Flashes (General disorders) | 1 (1)
Insomnia (General disorders) | 4 (7)
Pain (General disorders) | 1 (2)
Photosensiivity (Eye disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Prutitus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
This study was stopped early due to concerns about the interaction between St. John's wort and tamoxifen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No